CLINICAL TRIAL: NCT04924114
Title: A Phase 1b, Randomized, Adaptive, Double-Blind, Placebo-Controlled, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of PT101 in Subjects With Active Ulcerative Colitis
Brief Title: A Study of MK-6194 (PT101) in Participants With Active Ulcerative Colitis (UC) (MK-6194-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6194-002; PT101-201 (Other: Pandion); 2021-000093-28 (EudraCT Number)
Record Dates: First submitted 2021-02-26; First posted 2021-06-11 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MK-6194 Low Dose - Interval 1 (Less Frequent) (Experimental): Participants received low dose of MK-6194 at specified less frequent intervals
  Interventions: Drug: MK-6194
- MK-6194 Medium Dose- Interval 2 (More Frequent) (Experimental): Participants received medium dose of MK-6194 at specified more frequent intervals
  Interventions: Drug: MK-6194
- MK-6194 High Dose- Interval 2 (More Frequent) (Experimental): Participants received high dose of MK-6194 at specified more frequent intervals
  Interventions: Drug: MK-6194
- MK-6194 High Dose- Interval 1 (Less Frequent) (Experimental): Participants received high dose MK-6194 at specified less frequent intervals
  Interventions: Drug: MK-6194
- Placebo (Placebo Comparator): Participants received MK- 6194-matching placebo via subcutaneous injection, administered either at interval 1 or interval 2
  Interventions: Drug: MK-6194-matching placebo

INTERVENTIONS:
Drug: MK-6194 — Subcutaneous injection
  Other Names: PT101
  Arms: MK-6194 High Dose- Interval 1 (Less Frequent); MK-6194 High Dose- Interval 2 (More Frequent); MK-6194 Low Dose - Interval 1 (Less Frequent); MK-6194 Medium Dose- Interval 2 (More Frequent)
Drug: MK-6194-matching placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of MK-6194 in participants with active UC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC at least 3 months prior to screening.
* Mildly to severely active UC.
* Inadequate response, loss of response, or intolerance to at least 1 prior conventional therapy, and no more than 2 prior advanced therapies.
* Participants at risk for colorectal cancer must have a colonoscopy prior to or at screening as follows:

  * Participants > 50 years of age must have documentation of a colonoscopy within 3 years of the screening visit to exclude adenomatous polyps. Participants whose adenomas have been completely excised at screening are eligible.
  * Participants with extensive colitis for ≥ 8 years, or disease limited to the left side of the colon for ≥ 10 years, must either have had a full colonoscopy to assess for the presence of dysplasia within 1 year before first administration of study drug or a full colonoscopy to assess for the presence of malignancy at the screening visit.
* No evidence of active tuberculosis (TB), latent TB, or inadequately treated TB.
* Women of childbearing potential (WOCBP) and males with female partners of childbearing potential must utilize highly effective contraceptive methods beginning 4 weeks prior to first dose of study drug and continue for 30 days after the last dose of study drug.
* Body mass index (BMI) 18 to 35 kg/m^2 inclusive and weight ≥ 50 kg.

Exclusion Criteria:

* Prior treatment with recombinant IL-2 or modified IL-2 therapy, including MK-6194 (PT101).
* Known sensitivity to MK-6194 (PT101) or its excipients.
* Known history of hypersensitivity to interleukin-2 (IL-2).
* Disease limited to the rectum (i.e., within 15 cm of the anal verge).
* Diagnosis of toxic megacolon.
* Suspected or known colon stricture or stenosis.
* Diagnosis of Crohn's disease, or indeterminant colitis.
* Has severe colitis as evidenced by:

  * Current hospitalization for the treatment of UC
  * Likely to require a colectomy within 12 weeks of baseline in the opinion of the Investigator
  * At least 4 symptoms of severe colitis as identified at screening or baseline visits.
* Previously had surgery for UC, or likely to require surgery for UC during the study period in the opinion of the Investigator.
* History of abnormal thallium stress test or functional cardiac function test.
* History of significant cardiac, pulmonary, renal, hepatic, or central nervous system (CNS) impairment.
* Active clinically significant infection, or any infection requiring hospitalization or treatment with intravenous anti-infectives within 8 weeks of randomization, or any infection requiring oral anti-infective therapy within 6 weeks of randomization.
* History of opportunistic infection.
* History of symptomatic herpes zoster within 16 weeks of randomization, or any history of disseminated herpes simplex, disseminated herpes zoster, ophthalmic zoster, or central nervous system (CNS) zoster.
* Currently on any chronic systemic (oral or IV) anti-infective therapy for chronic infection (such as pneumocystis, cytomegalovirus, herpes zoster, or atypical mycobacteria).
* Currently receiving lymphocyte depleting therapy.
* History of abnormal pulmonary function tests.
* Participants with organ or tissue allograft.
* Malignancy within 5 years of screening, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin.
* Exposure to advanced therapy within 5 half-lives of the Day 1 visit, or documentation of detectable drug during screening.
* Received a live attenuated vaccine < 1 month prior to screening or is planning to receive a live attenuated vaccine during the study period or within 12 weeks of the end of participation in the study.
* Is pregnant or nursing or is planning to become pregnant during the study.
* Any uncontrolled or clinically significant concurrent systemic disease other than UC.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (17):
- United States (5):
  - Inland Empire Clinical Trials, LLC ( Site 0102), Rialto, California
  - IHS. Health, LLC ( Site 0104), Kissimmee, Florida
  - Carolina's GI Research, LLC ( Site 0105), Raleigh, North Carolina
  - Pinnacle Clinical Research ( Site 0103), San Antonio, Texas
  - Southern Star Research Institute ( Site 0101), San Antonio, Texas
- ARENSIA Exploratory Medicine Georgia ( Site 0801), Tbilisi, Georgia
- Charite Research Organisation GmbH ( Site 0201), Berlin, Germany
- PRA Magyarorszag Kutatasi es Fejlesztesi Kft. ( Site 0302), Budapest, Hungary
- ARENSIA Exploratory Medicine ( Site 0401), Chisinau, Moldova
- Poland (2):
  - Allmedica Badania Kliniczne Sp z o. o. Sp. K. ( Site 0502), Nowy Targ, Lesser Poland Voivodeship
  - WIP Warsaw IBD Point Professor Kierkus ( Site 0501), Warsaw, Masovian Voivodeship
- Arensia Exploratory Medicine GmbH Ukraine ( Site 0701), Kyiv, Kyivska Oblast, Ukraine
- United Kingdom (5):
  - MAC Clinical Research Prescot ( Site 0604), Prescot, Knowsley
  - Memory Assessment Clinics Ltd ( Site 0601), Blackpool, Lancashire
  - MAC Clinical Research ( Site 0602), Barnsley
  - MAC Clinical Research Centre Leeds ( Site 0603), Leeds
  - MAC Clinical Research Ltd. ( Site 0605), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26658&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon concluding the Initial Blinded Treatment (IBT) phase, participants could either complete the study or enter one of the next 2 phases. Participants who achieved clinical response could enter the continued blinded treatment (CBT) phase and continue receiving the same treatment as the IBT phase. Participants who did not achieve clinical response could enter an open label (OL) phase and receive MK-6194 at the same dose/regimen of their IBT cohort for active MK-6194 treatment.
Groups:
- MK-6194 High Dose - Interval 2 (More Frequent): Participants received high dose of MK-6194 at specified more frequent intervals
- MK-6194 High Dose - Interval 1 (Less Frequent): Participants received high dose MK-6194 at specified less frequent intervals
- Placebo: Participants received MK-6194-matching placebo via subcutaneous injection, administered either at interval 1 or interval 2
Period: Overall Study
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Started (All participants started in the IBT phase) | 7 | 11 | 18 | 10 | 11
Continued in CBT Phase (Participants who achieved clinical response after IBT phase could enter the continued blinded treatment (CBT) phase and continue receiving the same treatment as the IBT phase.) | 2 | 1 | 2 | 3 | 3
Treated in CBT Phase | 2 | 1 | 2 | 3 | 3
Continued in OL Phase (Participants who did not achieve clinical response after IBT phase could enter an open label (OL) phase and receive MK-6194 at the same dose/regimen of their IBT cohort for active MK-6194 treatment.) | 2 | 3 | 4 | 0 | 2
Treated in OL Phase (2 participants who received placebo in IBT phase received MK-6194 at the same dose/regimen of their IBT cohort for active MK-6194 treatment) | 3 (1 participant who received placebo in IBT phase received MK-6194 1mg Q4W in the OL phase) | 4 (1 participant who received placebo in IBT phase received MK-6194 2.5mg Q2W in the OL phase) | 4 | 0 | 0
Completed | 7 | 9 | 16 | 10 | 9
Not Completed | 0 | 2 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo | Total
Number analyzed (Participants) | 7 | 11 | 18 | 10 | 11 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (11.59) | 43.4 (14.64) | 47.7 (11.43) | 43.3 (10.11) | 35.6 (11.85) | 43.2 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 7 | 3 | 5 | 24
  Male | 3 | 6 | 11 | 7 | 6 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 3 | 5
  Not Hispanic or Latino | 5 | 11 | 18 | 9 | 8 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1 | 2
  White | 7 | 10 | 18 | 10 | 10 | 55
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Maximum Concentration (Cmax) of MK-6194
Description: Blood samples were collected at pre-specified time points to determine each participant's maximum concentration (Cmax). A participant's Cmax was defined as the maximum concentration of MK-6194 observed in serum over the entire course of the study for that individual and was calculated by taking the maximum over all observed MK-6194 serum concentrations. Geometric mean and geometric coefficient of variation of Cmax were calculated for each dosing group.
Time Frame: Predose on all days of dosing; 12, 24-48, and 120 hours (as available) post dose on the first and last day of dosing; and once each week up to approximately day 85.
Population: All randomized participants who received at least 1 dose of study intervention and who had least 1 valid analytical result at baseline, at least 1 post-dose analytical result and had no major relevant protocol or dosing deviations that could potentially affect the pharmacokinetic (PK) profile. Per protocol, samples from participants who received placebo were not analyzed for PK values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- MK-6194 Low Dose - Interval 1 (Less Frequent): Participants received low dose of MK-6194 at specified less frequent intervals test
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 7 | 9 | 18 | 10 | 0
ng/mL | 9.55 (67.80) | 30.02 (95.85) | 51.80 (71.97) | 52.78 (178.96) |

2. Secondary Outcome: Time to Cmax (Tmax) of MK-6194
Description: Blood samples were collected at pre-specified time points to determine maximum concentration (Cmax) of MK-6194 in each participant's serum and corresponding time of maximum concentration (Tmax). A participant's Tmax was defined as the time post-dose that the maximum concentration of MK-6194 was observed in serum. The median and range of Tmax were calculated for each dosing group.
Time Frame: as for outcome 1
Population: All randomized participants who received at least 1 dose of study intervention and who had least 1 valid analytical result at baseline, at least 1 post-dose analytical result and had no major relevant protocol or dosing deviations that could potentially affect he pharmacokinetic (PK) profile. Per protocol, samples from participants receiving placebo were not analyzed for PK values.
Measure: Median (Full Range); unit: hours
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 7 | 9 | 18 | 10 | 0
hours | 12.00 [11.10 to 24.00] | 12.00 [11.50 to 24.50] | 12.05 [11.10 to 25.00] | 12.10 [11.20 to 12.20] |

3. Secondary Outcome: Minimum Concentration (Cmin) of MK-6194
Description: Blood samples were collected at pre-specified time points to determine the minimum concentration (Cmin) of MK-6194 present in each participant's serum. A participant's Cmin was defined as the minimum concentration of MK-6194 observed in serum over the entire course of the study for that individual and was calculated by taking the minimum over all observed MK-6194 serum concentrations. Geometric mean and geometric coefficient of variation of Cmin were calculated for each dosing group.
Time Frame: as for outcome 1
Population: All randomized participants who received at least 1 dose of study intervention and who had least 1 valid analytical result at baseline, at least 1 post-dose analytical result and had no major relevant protocol or dosing deviations that could potentially affect the PK profile. Per protocol, samples participants receiving placebo were not analyzed for PK values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 7 | 9 | 18 | 10 | 0
ng/mL | 0.08 (0.00) | 0.08 (0.00) | 0.09 (97.70) | 0.08 (0.00) |

4. Secondary Outcome: Apparent Half-life (t1/2) of MK-6194
Description: Blood samples were collected at pre-specified time points to determine the apparent half-life (t1/2) of MK-6194. Noncompartmental analysis was used to calculate t1/2 for each participant using the terminal elimination phase after the final dose. Geometric mean and geometric coefficient of variation of t1/2 were calculated for each dosing group.
Time Frame: Final day of dosing at 12, 24-48 hours, and 120 hours (as available) post-dose; from the last day of dosing once each week up to approximately day 85
Population: All randomized participants who received at least 1 dose of study intervention and who had least 1 valid analytical result at baseline, at least 1 post-dose analytical result and had no major relevant protocol or dosing deviations that could potentially affect the PK profile. Per protocol, samples from participants receiving placebo were not analyzed for PK values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 6 | 5 | 10 | 9 | 0
hours | 193.28 (66.51) | 52.84 (23.89) | 42.06 (80.41) | 96.09 (16.51) |

5. Secondary Outcome: Apparent Clearance (CL/F) of MK-6194
Description: Blood samples were collected at pre-specified time points to determine the apparent clearance (CL/F) of MK-6194 observed in serum. Noncompartmental analysis was used to calculate CL/F for each participant using the terminal elimination phase after the final dose. Geometric mean and geometric coefficient of variation of CL/F were calculated for each dosing group.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hours
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 7 | 9 | 18 | 10 | 0
L/hours | 0.00 (66.28) | 0.01 (82.72) | 0.01 (95.07) | 0.01 (78.70) |

6. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of MK-6194
Description: Blood samples were collected at pre-specified time points to determine the apparent volume of distribution (Vd/F) of MK-6194 observed in serum. Noncompartmental analysis was used to calculate Vd/F for each participant using the terminal elimination phase after the final dose. Geometric mean and geometric coefficient of variation of Vd/F were calculated for each dosing group.
Time Frame: as for outcome 4
Population: All randomized participants who received at least 1 dose of study intervention and who had least 1 valid analytical result at baseline, at least 1 post-dose analytical result and had no major relevant protocol or dosing deviations that could potentially affect the PK profile. Per protocol, samples from participants who received placebo were not analyzed for PK values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 6 | 5 | 10 | 9 | 0
Liters | 1.61 (121.12) | 0.82 (96.99) | 0.55 (226.96) | 0.81 (93.17) |

7. Secondary Outcome: Area Under the Concentration Time-curve From Time 0 to the Last Quantifiable Concentration (AUC0-t)
Description: Blood samples were collected at pre-specified timepoints to determine the AUC0-t of MK-6194. AUC0-t is defined as the area under the concentration-time curve from time=0 (Day 1 predose) to the last quantifiable concentration. Noncompartmental analysis was used to calculate AUC0-t for each participant. Geometric mean and geometric coefficient of variation of AUC0-t were calculated for each dosing group.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 7 | 9 | 18 | 10 | 0
ng*hour/mL | 955.51 (39.92) | 2080.46 (55.64) | 3546.54 (67.17) | 3203.50 (117.92) |

8. Secondary Outcome: Area Under the Curve From Time 0 to Infinity (AUC0-inf) of MK-6194
Description: Blood samples were collected at pre-specified timepoints to determine the AUC0-inf of MK-6194. AUC0-inf is defined as the area under the concentration-time curve from time=0 (Day 1 predose) to time=infinity. Noncompartmental analysis was used to calculate AUC0-inf for each participant; the portion of the AUC following the last observed concentration was assumed to follow an exponential elimination. Geometric mean and geometric coefficient of variation of AUC0-inf were calculated for each dosing group.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 6 | 5 | 10 | 9 | 0
ng*hour/mL | 899.08 (36.53) | 2036.51 (71.46) | 3437.33 (65.59) | 3169.11 (120.37) |

9. Secondary Outcome: Change in Number of Peripheral Regulatory T-cells (Tregs) in Whole Blood
Description: Blood samples were collected at pre-specified time points and analyzed by flow cytometry. The absolute change in the number of peripheral Tregs in whole blood was assessed.
Time Frame: Pre-dose (baseline) and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: All randomized participants who received at least 1 dose of study intervention and who had least 1 valid analytical result at baseline, at least 1 post-dose analytical result and had no major relevant protocol or dosing deviations that could potentially affect the pharmacodynamic profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Cells/uL
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 3 | 11 | 18 | 10 | 9
Cells/uL
  Week 1: number analyzed (Participants) | 3 | 10 | 18 | 10 | 8
  Week 1 | 16.6 (46.10) | 24.0 (130.34) | 36.5 (76.68) | 31.0 (48.95) | 0.0 (107.20)
  Week 2: number analyzed (Participants) | 3 | 9 | 17 | 10 | 8
  Week 2 | 15.2 (45.43) | 8.4 (78.56) | 0.0 (84.52) | 29.8 (100.53) | 6.0 (109.31)
  Week 3: number analyzed (Participants) | 2 | 10 | 16 | 10 | 8
  Week 3 | 12.2 (113.83) | 24.5 (95.40) | 31.7 (92.24) | 15.2 (77.36) | 4.4 (96.26)
  Week 4: number analyzed (Participants) | 3 | 9 | 16 | 9 | 7
  Week 4 | 5.1 (71.20) | 9.5 (78.31) | 12.8 (82.29) | 4.8 (115.02) | 0.0 (120.87)
  Week 5: number analyzed (Participants) | 3 | 8 | 14 | 10 | 9
  Week 5 | 33.9 (61.55) | 0.0 (66.63) | 20.9 (78.63) | 35.5 (65.56) | 0.0 (92.71)
  Week 6: number analyzed (Participants) | 3 | 8 | 15 | 7 | 6
  Week 6 | 9.0 (32.73) | 12.9 (73.27) | 9.8 (100.16) | 18.9 (58.45) | 0.0 (61.81)
  Week 7: number analyzed (Participants) | 3 | 5 | 14 | 9 | 7
  Week 7 | 4.0 (53.29) | 32.3 (44.51) | 27.1 (69.98) | 7.4 (130.11) | 0.0 (66.82)
  Week 8: number analyzed (Participants) | 3 | 6 | 13 | 9 | 8
  Week 8 | 3.9 (25.00) | 9.4 (101.40) | 8.8 (62.20) | 7.7 (101.49) | 0.0 (102.85)
  Week 9: number analyzed (Participants) | 3 | 5 | 14 | 9 | 8
  Week 9 | 6.0 (121.24) | 21.1 (76.45) | 22.3 (83.28) | 42.1 (63.99) | 4.3 (101.64)
  Week 10: number analyzed (Participants) | 3 | 8 | 13 | 9 | 7
  Week 10 | 2.3 (24.74) | 15.4 (55.42) | 11.3 (76.11) | 16.3 (91.23) | 3.5 (146.88)
  Week 11: number analyzed (Participants) | 0 | 8 | 12 | 0 | 5
  Week 11 |  | 17.8 (79.90) | 24.6 (82.30) |  | 3.5 (117.48)
  Week 12: number analyzed (Participants) | 3 | 8 | 13 | 9 | 8
  Week 12 | 5.9 (16.67) | 12.1 (56.51) | 6.4 (89.54) | 0.0 (77.22) | 4.7 (91.20)

10. Secondary Outcome: Change in Number of Natural Killer (NK) Cells in Whole Blood
Description: Blood samples were collected at pre-specified time points and analyzed by flow cytometry. The change in the number of NK cells in whole blood is presented.
Time Frame: Pre-dose (baseline) and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Cells/uL
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 3 | 11 | 18 | 10 | 9
Cells/uL
  Week 1: number analyzed (Participants) | 3 | 10 | 18 | 10 | 8
  Week 1 | 109.3 (117.56) | 0.0 (149.43) | 43.2 (86.39) | 110.0 (61.90) | 34.40 (60.38)
  Week 2: number analyzed (Participants) | 3 | 9 | 17 | 10 | 8
  Week 2 | 124.7 (83.32) | 76.1 (62.77) | 48.6 (81.20) | 108.5 (55.48) | 19.2 (160.68)
  Week 3: number analyzed (Participants) | 2 | 10 | 16 | 10 | 8
  Week 3 | 479.5 (85.51) | 50.3 (73.79) | 44.2 (110.61) | 68.4 (62.20) | 64.1 (87.37)
  Week 4: number analyzed (Participants) | 3 | 9 | 16 | 9 | 7
  Week 4 | 292.2 (48.38) | 52.8 (67.48) | 0.0 (102.83) | 78.9 (73.40) | 42.1 (131.09)
  Week 5: number analyzed (Participants) | 3 | 8 | 14 | 10 | 9
  Week 5 | 281.5 (27.43) | 42.1 (76.34) | 53.8 (61.16) | 133.2 (87.96) | 65.0 (129.61)
  Week 6: number analyzed (Participants) | 3 | 8 | 15 | 7 | 6
  Week 6 | 169.0 (88.11) | 59.3 (72.56) | 54.7 (80.71) | 140.3 (78.10) | 55.3 (124.75)
  Week 7: number analyzed (Participants) | 3 | 5 | 14 | 9 | 7
  Week 7 | 224.8 (83.09) | 0.0 (112.85) | 73.2 (66.16) | 82.0 (93.62) | 44.9 (119.10)
  Week 8: number analyzed (Participants) | 3 | 6 | 13 | 9 | 8
  Week 8 | 272.9 (54.62) | 38.4 (113.46) | 43.7 (148.37) | 86.9 (49.10) | 30.4 (125.05)
  Week 9: number analyzed (Participants) | 3 | 5 | 14 | 9 | 8
  Week 9 | 195.5 (4.35) | 92.8 (94.04) | 72.8 (74.20) | 94.0 (75.86) | 53.2 (81.75)
  Week 10: number analyzed (Participants) | 3 | 8 | 13 | 9 | 7
  Week 10 | 159.6 (59.86) | 26.4 (83.25) | 46.0 (111.12) | 87.1 (99.38) | 84.5 (91.34)
  Week 11: number analyzed (Participants) | 0 | 8 | 12 | 0 | 5
  Week 11 |  | 42.3 (94.19) | 47.0 (91.92) |  | 41.1 (163.74)
  Week 12: number analyzed (Participants) | 3 | 8 | 13 | 9 | 8
  Week 12 | 70.6 (125.61) | 67.6 (60.56) | 58.4 (84.39) | 45.6 (119.58) | 40.9 (121.60)

11. Secondary Outcome: Change in Number of Conventional T Cells (Tcons) in Whole Blood
Description: Blood samples were collected at pre-specified time points and analyzed by flow cytometry. The change in the number of Tcons in whole blood is presented.
Time Frame: Pre-dose (baseline) and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Cells/uL
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 3 | 11 | 18 | 10 | 9
Cells/uL
  Week 1: number analyzed (Participants) | 3 | 10 | 18 | 10 | 8
  Week 1 | 216.9 (94.52) | 220.8 (94.37) | 91.2 (105.12) | 189.6 (66.58) | 57.6 (79.00)
  Week 2: number analyzed (Participants) | 3 | 9 | 17 | 10 | 8
  Week 2 | 106.1 (124.15) | 100.8 (67.50) | 105.4 (121.23) | 184.1 (67.77) | 0.0 (71.58)
  Week 3: number analyzed (Participants) | 2 | 10 | 16 | 10 | 8
  Week 3 | 347.3 (129.76) | 81.1 (98.95) | 123.7 (111.06) | 192.8 (60.55) | 127.7 (52.96)
  Week 4: number analyzed (Participants) | 3 | 9 | 16 | 9 | 7
  Week 4 | 280.2 (116.12) | 122.4 (61.71) | 73.3 (108.47) | 163.4 (72.06) | 63.3 (105.58)
  Week 5: number analyzed (Participants) | 3 | 8 | 14 | 10 | 9
  Week 5 | 456.3 (28.23) | 100.6 (74.36) | 126.2 (75.69) | 166.8 (76.19) | 79.3 (66.49)
  Week 6: number analyzed (Participants) | 3 | 8 | 15 | 7 | 6
  Week 6 | 114.3 (119.18) | 57.9 (101.25) | 0.0 (101.48) | 193.9 (68.59) | 53.8 (90.84)
  Week 7: number analyzed (Participants) | 3 | 5 | 14 | 9 | 7
  Week 7 | 137.7 (84.27) | 103.6 (68.22) | 68.6 (87.88) | 154.5 (70.64) | 66.1 (87.17)
  Week 8: number analyzed (Participants) | 3 | 6 | 13 | 9 | 8
  Week 8 | 381.1 (34.64) | 109.0 (84.28) | 63.5 (82.18) | 159.1 (66.12) | 50.6 (93.80)
  Week 9: number analyzed (Participants) | 3 | 5 | 14 | 9 | 8
  Week 9 | 250.3 (39.38) | 164.1 (51.01) | 128.8 (89.61) | 192.2 (71.43) | 141.5 (63.25)
  Week 10: number analyzed (Participants) | 3 | 8 | 13 | 9 | 7
  Week 10 | 271.1 (81.50) | 33.4 (115.44) | 50.7 (98.06) | 147.3 (72.31) | 83.2 (92.61)
  Week 11: number analyzed (Participants) | 0 | 8 | 12 | 0 | 5
  Week 11 |  | 76.1 (59.20) | 90.5 (80.69) |  | 102.0 (45.66)
  Week 12: number analyzed (Participants) | 3 | 8 | 13 | 9 | 8
  Week 12 | 122.6 (134.20) | 73.2 (96.94) | 99.9 (77.32) | 153.3 (70.03) | 73.4 (82.45)

12. Secondary Outcome: Titer of Anti-drug Antibody (ADA) to MK-6194
Description: Blood samples were collected for the determination of ADA to MK-6194 using a screening assay, ADA titer using a confirmatory assay, and neutralizing antibody to MK-6194 in participants with confirmed positive titers
Time Frame: Pre dose (week 0) and Weeks 4, 8, 12
Population: All randomized participants who received at least 1 dose of study intervention and who had least 1 valid analytical result at baseline, at least 1 post-dose analytical result and had no major relevant protocol or dosing deviations that could potentially affect the pharmacodynamic profile. ADA titer was assessed only in participants who were ADA positive.
Measure: Median (Full Range); unit: Titer
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 1 | 5 | 8 | 7 | 0
Titer
  Week 0: number analyzed (Participants) | 0 | 1 | 0 | 2 | 0
  Week 0 |  | 20.0 [20.0 to 20.0] |  | 20.0 [20.0 to 20.0] |
  Week 4: number analyzed (Participants) | 0 | 3 | 3 | 4 | 0
  Week 4 |  | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 160.0] |
  Week 8: number analyzed (Participants) | 1 | 1 | 2 | 5 | 0
  Week 8 | 160.0 [160.0 to 160.0] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 40.0] |
  Week 12: number analyzed (Participants) | 1 | 3 | 6 | 6 | 0
  Week 12 | 640.0 [640.0 to 640.0] | 40.0 [20.0 to 320.0] | 20.0 [20.0 to 640.0] | 40.0 [20.0 to 160.0] |

13. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to approximately 85 days
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 7 | 11 | 18 | 10 | 11
Participants | 7 | 10 | 18 | 10 | 7

14. Primary Outcome: Number of Participants Who Interrupted or Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to thestudy intervention
Time Frame: Up to approximately 72 days
Population: All participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | MK-6194 Low Dose - Interval 1 (Less Frequent) | MK-6194 Medium Dose- Interval 2 (More Frequent) | MK-6194 High Dose - Interval 2 (More Frequent) | MK-6194 High Dose - Interval 1 (Less Frequent) | Placebo
Number analyzed (Participants) | 7 | 11 | 18 | 10 | 11
Participants | 1 | 0 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to approximately 52 weeks
Description: The population consists of all participants who received at least one dose of study drug. Treatment groups use the actual treatment received, regardless of randomization assignment. Per protocol, participants receiving placebo in IBT phase and not achieving clinical response could enter the OL phase to receive the matching MK-6194 regimen from their IBT cohort. Participants receiving placebo in IBT phase and achieving clinical response could enter the CBT phase and continue receiving placebo.
Groups:
- IBT: MK-6194 Low Dose Interval 1 (Less Frequent): Participants received low dose MK-6194 at specified less frequent intervals for up to 12 weeks
- IBT-MK-6194 Medium Dose- Interval 2 (More Frequent): Participants received medium dose of MK-6194 at specified more frequent intervals for up to 12 weeks
- IBT: MK-6194 High Dose-Interval 2 (More Frequent): Participants received high dose of MK-6194 at specified more frequent intervals for up to 12 weeks
- IBT:MK-6194 High Dose-Interval 1 (Less Frequent): Participants received high dose MK-6194 at specified less frequent intervals for up to 12 weeks
- IBT: Placebo: Participants received MK-6194-matching placebo via subcutaneous injection, administered either at interval 1 or interval 2 for up to 12 weeks
- CBT: MK-6194 Low Dose- Interval 1 (Less Frequent): Participants who achieved clinical response at week 12 of the IBT continued to receive low dose MK-6194 at specified less frequent intervals for up to 9 months
- CBT: MK-6194 Medium Dose- Interval 2 (More Frequent): Participants who achieved clinical response at week 12 of the IBT continued to receive medium dose MK-6194 at specified more frequent intervals for up to 9 months
- CBT: MK-6194 High Dose- Interval 2 (More Frequent): Participants who achieved clinical response at week 12 of the IBT continued to receive high dose MK-6194 at specified more frequent intervals for up to 9 months
- CBT: MK-6194 High Dose - Interval 1 (Less Frequent): Participants who achieved clinical response at week 12 of the IBT continued to receive high dose MK-6194 at specified less frequent intervals for up to 9 months
- CBT: Placebo: Participants who achieved clinical response at week 12 of the IBT continued to receive placebo at interval 1 or 2 for up to 9 months
- OL: MK-6194 Low Dose -Interval 1 (Less Frequent): Participants who did not achieve clinical response at week 12 received low dose MK-6194 at specified less frequent intervals for up to 9 months
- OL: MK-6194 Medium Dose- Interval 2 (More Frequent): Participants who did not achieve clinical response at week 12 received medium dose MK-6194 at specified more frequent intervals for up to 9 months
- OL: MK-6194 High Dose- Interval 2 (More Frequent): Participants who did not achieve clinical response at week 12 received high dose MK-6194 at specified more frequent intervals for up to 9 months
Arm/Group | IBT: MK-6194 Low Dose Interval 1 (Less Frequent) | IBT-MK-6194 Medium Dose- Interval 2 (More Frequent) | IBT: MK-6194 High Dose-Interval 2 (More Frequent) | IBT:MK-6194 High Dose-Interval 1 (Less Frequent) | IBT: Placebo | CBT: MK-6194 Low Dose- Interval 1 (Less Frequent) | CBT: MK-6194 Medium Dose- Interval 2 (More Frequent) | CBT: MK-6194 High Dose- Interval 2 (More Frequent) | CBT: MK-6194 High Dose - Interval 1 (Less Frequent) | CBT: Placebo | OL: MK-6194 Low Dose -Interval 1 (Less Frequent) | OL: MK-6194 Medium Dose- Interval 2 (More Frequent) | OL: MK-6194 High Dose- Interval 2 (More Frequent)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/11 | 0/18 | 0/10 | 0/11 | 0/2 | 0/1 | 0/2 | 0/3 | 0/3 | 0/3 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/11 | 1/18 | 0/10 | 0/11 | 0/2 | 0/1 | 0/2 | 0/3 | 0/3 | 0/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 7/7 | 10/11 | 18/18 | 10/10 | 7/11 | 2/2 | 1/1 | 2/2 | 2/3 | 1/3 | 1/3 | 3/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBT: MK-6194 Low Dose Interval 1 (Less Frequent) (N=7) | IBT-MK-6194 Medium Dose- Interval 2 (More Frequent) (N=11) | IBT: MK-6194 High Dose-Interval 2 (More Frequent) (N=18) | IBT:MK-6194 High Dose-Interval 1 (Less Frequent) (N=10) | IBT: Placebo (N=11) | CBT: MK-6194 Low Dose- Interval 1 (Less Frequent) (N=2) | CBT: MK-6194 Medium Dose- Interval 2 (More Frequent) (N=1) | CBT: MK-6194 High Dose- Interval 2 (More Frequent) (N=2) | CBT: MK-6194 High Dose - Interval 1 (Less Frequent) (N=3) | CBT: Placebo (N=3) | OL: MK-6194 Low Dose -Interval 1 (Less Frequent) (N=3) | OL: MK-6194 Medium Dose- Interval 2 (More Frequent) (N=4) | OL: MK-6194 High Dose- Interval 2 (More Frequent) (N=4)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBT: MK-6194 Low Dose Interval 1 (Less Frequent) (N=7) | IBT-MK-6194 Medium Dose- Interval 2 (More Frequent) (N=11) | IBT: MK-6194 High Dose-Interval 2 (More Frequent) (N=18) | IBT:MK-6194 High Dose-Interval 1 (Less Frequent) (N=10) | IBT: Placebo (N=11) | CBT: MK-6194 Low Dose- Interval 1 (Less Frequent) (N=2) | CBT: MK-6194 Medium Dose- Interval 2 (More Frequent) (N=1) | CBT: MK-6194 High Dose- Interval 2 (More Frequent) (N=2) | CBT: MK-6194 High Dose - Interval 1 (Less Frequent) (N=3) | CBT: Placebo (N=3) | OL: MK-6194 Low Dose -Interval 1 (Less Frequent) (N=3) | OL: MK-6194 Medium Dose- Interval 2 (More Frequent) (N=4) | OL: MK-6194 High Dose- Interval 2 (More Frequent) (N=4)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 3 (4) | 7 (26) | 17 (50) | 4 (8) | 2 (2) | 1 (2) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 1 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 5 (13) | 7 (19) | 12 (39) | 5 (8) | 0 (0) | 2 (5) | 1 (1) | 2 (6) | 1 (5) | 0 (0) | 1 (3) | 2 (5) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 2 (4) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatillomania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator will submit the proposed publication to the sponsor at least 30 days prior to the date of submission for publication. The sponsor can request to remove any confidential information other than study data from a proposed publication during the review period. The sponsor may also suggest changes to the presentation of study data and timing of the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT04924114/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT04924114/SAP_001.pdf